CLINICAL TRIAL: NCT01545167
Title: The North American Pancreatitis Study
Acronym: NAPS
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, David Whitcomb, Chief, Division of Gastroenterology, Hepatology and Nutrition, University of Pittsburgh
Other Study IDs: DK 061451; NAPS2-AS (Other Grant/Funding Number: R01 DK077906)
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Pancreatitis
Keywords: African Americans; pancreatitis; controls
MeSH Terms: conditions — Pancreatitis | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples and extracted biomarkers and genetic material.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- African Americans with pancreatitis: pancreatitis
  Interventions: Genetic: blood sampling
- African Americans without Pancreatitis controls: people without pancreatitis
  Interventions: Genetic: blood sampling

INTERVENTIONS:
Genetic: blood sampling — blood samples obtained to extract biomarkers and dna for analysis, questionnaires

SUMMARY:
This study will investigate several genes and other factors measured in the blood that may cause recurrent acute pancreatitis and chronic pancreatitis. No treatment is offered as part of this study. Subjects have one single visit to provide a blood sample for genetic testing and to answer a questionnaire. Subjects are not given results of genetic testing. The study is currently enrolling African American subjects and controls only.

DETAILED DESCRIPTION:
This study seeks to enroll African American people with and without pancreatitis. There is only one study visit to obtain consent, a blood sample and complete a questionnaire. Subjects must be patients of a participating center; controls must present to a participating center for enrollment.

ELIGIBILITY:
Inclusion Criteria:

African American

pancreatitis patients who are at least 14 years of age with a diagnosis of acute or chronic pancreatitis

* controls who do not have pancreatitis and must be at least 18 years of age

Exclusion Criteria:

* unable or unwilling to sign informed consent

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: people with and without pancreatitis
Sampling Method: Non-Probability Sample
Enrollment: 2980 (Actual)
Dates: Start 2008-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Yadav D, Whitcomb DC, Tang G, Slivka A, Bellin M; North American Pancreatitis Studies Consortium. Autoimmunity May Explain Diabetes in a Subset of Patients With Recurrent Acute and Chronic Pancreatitis: A Pilot Study. Clin Gastroenterol Hepatol. 2023 Jan;21(1):226-228.e1. doi: 10.1016/j.cgh.2021.11.011. Epub 2021 Nov 16. PMID 34793964
- [Derived] Dunbar EK, Greer PJ, Amann ST, Alkaade S, Banks P, Brand R, Conwell DL, Forsmark CE, Gardner TB, Guda NM, Lewis MD, Machicado JD, Muniraj T, Papachristou GI, Romagnuolo J, Sandhu BS, Sherman S, Slivka A, Wilcox CM, Yadav D, Whitcomb DC; NAPS2 Consortium. Pain Experience in Pancreatitis: Strong Association of Genetic Risk Loci for Anxiety and PTSD in Patients With Severe, Constant, and Constant-Severe Pain. Am J Gastroenterol. 2021 Oct 1;116(10):2128-2136. doi: 10.14309/ajg.0000000000001366. PMID 34236339
- [Derived] Dunbar E, Greer PJ, Melhem N, Alkaade S, Amann ST, Brand R, Cote GA, Forsmark CE, Gardner TB, Gelrud A, Guda NM, LaRusch J, Lewis MD, Machicado JD, Muniraj T, Papachristou GI, Romagnuolo J, Sandhu BS, Sherman S, Wilcox CM, Singh VK, Yadav D, Whitcomb DC; NAPS2 study group. Constant-severe pain in chronic pancreatitis is associated with genetic loci for major depression in the NAPS2 cohort. J Gastroenterol. 2020 Oct;55(10):1000-1009. doi: 10.1007/s00535-020-01703-w. Epub 2020 Jul 17. PMID 32681239